CLINICAL TRIAL: NCT05446922
Title: National, Multicentre, Prospective, Interventional Study of the Variability of Cerebral MRI Diffusion Parameters by Using a Patented Normalization Process Versus no Use of Normalization Process
Brief Title: Variability of Cerebral MRI Diffusion Parameters by Using a Patented Normalization Process vs no Use
Acronym: CALI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Braintale (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00622-41
Record Dates: First submitted 2022-06-15; First posted 2022-07-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Brain MRI
MeSH Terms: interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI imaging of 10 healthy volunteers (Other): 10 healthy volunteers will proceed at an brain MRI imaging
  Interventions: Other: Diffusion MRI

INTERVENTIONS:
Other: Diffusion MRI — All procedures will be performed during a single visit. Subjects will be invited to lie on the scanning bed that will be moved head first into the scanner such as the head lie under the scanner magnets. Hearing protection will be provided to each subject to muffle the noise produced by the MRI scanner. Subjects will also be provided with pillows and blankets to keep them comfortable. They will also be given a call button that they can push to stop the procedure at any time. MRI acquisition will be performed on 1.5T or 3.0T MRI scanners depending on centre's equipment. Acquisition protocol will include the following sequences with the best parameters chosen by local radiologist and technical BrainTale team.

SUMMARY:
BrainTale has developed a standardization approach based on averaging measurements in predefined brain regions of interest and use of reference data acquired from healthy volunteers under conditions (MRI machine, acquisition protocol) identical to those used for the examination of the patient. The present study is intended to support the normalization step on healthy volunteers in clinical centres that will be equipped with the BrainTale medical device software dedicated to clinical routine practice and to assess, through a multicentre study, the impact of this normalization step on the variability of the MRI diffusion parameters. The data collected will support characterization and modelisation of the variability to explore further biais corrections methods. The study will be conducted by neuroradiologists of the neuroradiology departments of five clinical centres in France.

DETAILED DESCRIPTION:
Advances in medical imaging have made it possible, from the 1990s, to be able to visualize structural microlesions of the brain thanks to post-processing of the Magnetic Resonance Imaging (MRI) data acquired by the sequence using the diffusion tensor. Mathematical models such as the diffusion tensor have made it possible to quantify in each of the volumetric units of the brain (voxels) measurements correlated to the microstructure of neuronal axons such as the Fractional Anisotropy (FA), the Mean Diffusivity (MD), the Radial Diffusivity (RD) or the Axial Diffusivity (AD). These measurements thus make it possible to quantify the microstructural alterations.

However, the use of Diffusion Tensor Imaging (DTI) technology has limitations and currently, there is no "gold-standard" to validate diffusion measurements, which are currently dependent on acquisition protocols, post-processing software and observers.

To make these diffusion parameters usable in a clinical context, BrainTale has developed a standardization approach based on averaging measurements in predefined brain regions of interest and use of reference data acquired from healthy volunteers under conditions (MRI machine, acquisition protocol) identical to those used for the examination of the patient. This process requires the acquisition of 10 healthy volunteers to calibrate a new MRI protocol, which greatly limits access to the technology in clinical routine and limits the potential technological evolutions of the acquisition.

The study aims to assess the impact of a patented normalization process on the interindividual variability of Fractional Anisotropy (FA) measurements derived from cerebral Diffusion Tensor Imaging (DTI) acquisitions.

A total of 60 healthy volunteers will be included. One or two acquisition will be performed during a single on-site visit in order to collect diffusion parameters outcome data for further analyses (with or without normalization process).

After each acquisition and before inclusion of the following healthy volunteer, anonymised subject's data will be transferred to BrainTale on a secured web platform. BrainTale will be in charge of the Quality Control (QC) of the acquired data and will attribute a QC-passed or QC-failed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 up to 80 years old
2. Covered by a healthcare insurance
3. Agreeing to be informed about any incidental finding discovered on brain MRI
4. Written informed consent form signed

Exclusion Criteria:

1. History of brain pathology, cognitive or psychiatric disorder
2. Any contraindication * for undergoing brain MRI
3. Subject refusing to participate or having expressed refusal to data collection/processing or unable to give his/her agreement to participate
4. Vulnerable subject (i.e. pregnant or breast-feeding woman, child, subject under curatorship or deprived of liberty)

   * contraindications to MRI include: pacemaker, neural stimulator, intraocular or intracerebral device, cochlear implant, MR-incompatible prosthetic heart valves, any implant with metallic, ferromagnetic or electrically conductive parts, any metal in the body which cannot be removed, claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Coefficients of Variation (%CV) of FA measurement | Day 1
  Percentage Coefficients of Variation (%CV) of FA measurements obtained from QC-passed DTI sequences before and after application of the normalization process.

SECONDARY OUTCOMES:
Coefficients of Variation (%CV) of MD measurement | Day 1
  Percentage Coefficients of Variation (%CV) of MD measurements obtained from QC-passed DTI sequences before and after application of the normalization process.
Coefficients of Variation (%CV) of AD measurement | Day 1
  Percentage Coefficients of Variation (%CV) of AD measurements obtained from QC-passed DTI sequences before and after application of the normalization process.
Coefficients of Variation (%CV) of RD measurement | Day 1
  Percentage Coefficients of Variation (%CV) of RD measurements obtained from QC-passed DTI sequences before and after application of the normalization process.

OTHER OUTCOMES:
Intraclass Correlation Coefficient (ICC) | Day 1
  For assessment of the impact of calibration on test-retest repeatability of cerebral MRI diffusion parameters.
  The Intraclass Correlation Coefficient (ICC) of cerebral MRI diffusion parameters (FA, MD, RD, AD) between the two measures made on the same patients, per center.
percentage Coefficient of Variation (%CV) of the Neurite Orientation Dispersion and Density Imaging (NODDI) multishell diffusion scalar parameters. | Day 1
  For assessment of the variability of multishell diffusion parameters:
  The percentage Coefficient of Variation (%CV) of the Neurite Orientation Dispersion and Density Imaging (NODDI) multishell diffusion scalar parameters, i.e. Neurite Density Index (NDI), Orientation Dispersion Index (ODI) and Free Water fraction (FW).
percentage Coefficient of Variation (%CV) of the resting-state functional MRI (fMRI) parameters. | Day 1
  For assessment of the variability of resting state fMRI parameters:
  The percentage Coefficient of Variation (%CV) of the resting-state functional MRI (fMRI) parameters: Regional Homogeneity (ReHo) and functional integration metrics.

CONTACTS AND LOCATIONS:
Overall Officials: PERLBARG Vincent, Study Chair — Braintale

IPD SHARING:
Plan to Share IPD: No